CLINICAL TRIAL: NCT02010242
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Study Evaluating the Safety and Efficacy of Oral GKT137831 in Patients With Type 2 Diabetes and Albuminuria
Brief Title: Safety and Efficacy of Oral GKT137831 in Patient With Type 2 Diabetes and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSN000200
Record Dates: First submitted 2013-06-18; First posted 2013-12-12 (Estimated); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus With Diabetic Nephropathy
Keywords: Type 2 diabetes; Proteinuria; Albuminuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria; Albuminuria | interventions — setanaxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GKT137831 (Experimental): GKT137831 100 mg capsules twice a day
  Interventions: Drug: GKT137831
- Placebo (Placebo Comparator): Placebo capsule twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GKT137831 — 1 capsule of 100 mg twice a day for the first 6 weeks of treatment, and 2 capsules of 100 mg twice a day for next 6 weeks of treatment
  Arms: GKT137831
Drug: Placebo — 1 capsule of Placebo, twice a day, oral treatment self-administered by the patient for the 12 weeks of treatment.
  Arms: Placebo

SUMMARY:
NADPH oxidase enzymes (NOX) have been implicated in the development of several diabetic complications including diabetic nephropathy. GKT137831 is the first in class NOX1/4 inhibitor.

The primary objective of this study is to evaluate the efficacy of oral GKT137831 in patients with residual albuminuria despite maximal inhibition of the renin angiotensin aldosterone system.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, randomized, multicenter, parallel group Phase 2 study assessing a 12-week period of treatment with oral GKT137831 administered in addition to standard of care for patients with type 2 diabetes.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged 18 to 80 years
* History of type 2 diabetes, defined as fasting plasma glucose ≥7.0 mmol/L (126 mg/dL) or a glycated hemoglobin (HbA1c) >6.5% (48 mmol/mol) on at least 2 occasions prior to screening.
* Albuminuria defined as a UACR of 300 to 3500 mg/g.
* An eGFR ≥30 mL/min/1.73 m2, as calculated by the CKD-EPI formula.
* Must be taking an ACEI or an ARB for at least 6 weeks prior to the first screening visit (Visit 1) and during the screening period. The dose must have been stable for at least 4 weeks prior to the first screening visit (Visit 1). Combination therapy associating an ACEI and an ARB is not permitted.

Key Exclusion Criteria:

* History of type 1 diabetes
* Any other non-diabetic kidney disease(s) except for hypertensive nephropathy which is acceptable.
* Diagnostic or interventional procedure requiring a contrast agent within 4 weeks of the first screening visit (Visit 1) or planned during the study.
* History of renal transplant or planned renal transplant during the study.
* A history of acute renal dialysis or acute kidney injury (defined according to the Kidney Disease: Improving Global Outcomes [KDIGO] definition) within 12 weeks of the first screening visit (Visit 1)
* HbA1c level >11% (97 mmol/mol).
* History of hypothyroidism requiring hormone replacement therapy.
* History of active cardiovascular disease
* A personal or family history of long QT syndrome.
* Administration of any investigational product within 30 days or within 5 half-lives of the investigational agent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Wiesel, MD, Study Director — Calliditas Therapeutics AB
Locations (48):
- United States (20):
  - Advanced Arizona Clinical Research, Tucson, Arizona
  - The Endocrine Medical Group, Inc, Orange, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Coral Research Clinic, Miami, Florida
  - Pines Clinical Research Inc., Pembroke Pines, Florida
  - Volunteer Medical Research, Port Charlotte, Florida
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Community Medical Research Partners, Indianapolis, Indiana
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Creighton Diabetes Center, Omaha, Nebraska
  - LLC DBA AccessMD Clinical Research, Dayton, Ohio
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - 17070 Red Oak dr Ste 103, Houston, Texas
  - Dialysis West University Health System, San Antonio, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - Zablocki VAMC, Milwaukee, Wisconsin
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Deakin University school of medicine, Geelong, Victoria
  - Austin Health, Heidelberg, Victoria
  - Baker Institute, Melbourne, Victoria
  - Maroondah ECRU, Ringwood East, Victoria
  - Captain Stirling Medical Centre, Nedlands, Western Australia
- Canada (6):
  - Endocrine Research Inc., Vancouver, British Columbia
  - LMC Diabetes & Endocrinology, Brampton, Ontario
  - Clinical Research Solutions, Kitchener, Ontario
  - LMC Diabetes and Endocrinology, Thornhill, Ontario
  - Toronto East General Medical Centre, Toronto, Ontario
  - Medpharmgene, Montreal, Quebec
- Czechia (5):
  - Nemocnice Havlickuv Brod, Huzová
  - Oblastni nemocnice Jicin a.s., Nový Bydžov
  - Faculty Hospital and Palacky University Olomouc, Olomouc
  - Milan Kvapil s.r.o. diabetology ambulance, Prague
  - IKEM, Prague
- Germany (4):
  - Studienzentrum Haematologie/Onkologie/Diabeteologie, Aschaffenburg
  - ZKS Suedbrandenburg GmbH, Elsterwerda
  - IKFE - Institute for Clinical Research and Development, Mainz
  - IDFM, München
- Poland (7):
  - Centrum Badaa Klinicznych PI-House Sp. z o.o., Gdansk
  - LANDA Specjalistyczne Gabinety Lekarskie, Krakow
  - Medicus w Opolu sp z o.o., Opole
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - KO-MED Centra Kliniczne Sp. z o.o., Staszów
  - Department of Nephrology, Transplantationa and Internal Medicine, Szczecin
  - Medica Pro Familia Sp. z o.o. S.K.A., Warsaw

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GKT137831 | Placebo
Started | 68 | 68
Completed | 64 | 61
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GKT137831 | Placebo | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 43 | 81
  >=65 years | 30 | 25 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (8.64) | 62.2 (9.9) | 62.1 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 52 | 52 | 104
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 9 | 21
  United States | 26 | 30 | 56
  Czechia | 13 | 8 | 21
  Poland | 5 | 8 | 13
  Australia | 5 | 11 | 16
  Germany | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Albuminuria Absolute Value and Ratio to Baseline by Study Visit and Treatment Group
Description: UACR from baseline to Visits 9, 10, and 11 (i.e. weeks 8, 10 and 12 of the treatment period, respectively).
  Baseline for UACR is defined as the geometric mean of the geometric means of the UACR values measured on Day-14 (visit 4) and Day 1 (visit 5). End of treatment is defined as the geometric mean of the geometric means of the UACR values measured at week 8 (visit 9), week 10 (visit 10) and week 12 (visit 11).
Time Frame: Visit 4 (week -2) to visit 11 (week 12)
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Geometric Mean (90% Confidence Interval); unit: mg/g
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 62 | 59
mg/g
  Baseline Geom. Mean | 705.72 [637.07 to 774.36] | 696.30 [611.98 to 780.61]
  Adjusted End of treatment Geom. Mean | 758.22 [695.61 to 826.46] | 705.29 [646.19 to 769.80]
Statistical Analysis 1: Comparison: GKT137831 vs Placebo; Primary efficacy endpoint was analyzed using ANCOVA comparing GKT137831 vs placebo after controlling for the baseline UACR level. The UACR were log-transformed prior to analysis. The model included treatment group and log-transformed baseline UACR value as predicted variables. The results were back-transformed exponentially to calculate geo. mean values and associated 90% CIs and 1-sided p-values. The null hypothesis was that the difference in the adjusted mean logarithm of UACR was equal to 0; Test type: Superiority — All statistical analyses were performed on a comparison-wise basis without adjustment for multiple comparisons; p = 1.000, ANCOVA

2. Secondary Outcome: Glucose Metabolism by Homeostatic Model Assessment (HOMA)
Description: Change in homeostasis model assessment-estimated β cell function (HOMA-B) and homeostasis model assessment-estimated insulin resistance (HOMA-IR) from baseline.
  HOMA-IR = fasting insulin (μIU/mL) x fasting glucose (mM/L)/22.5. A higher HOMA-IR value indicates greater insulin resistance.
  HOMA-B = 20 x fasting insulin (μIU/mL)/(fasting glucose [mmol/mL] - 3.5). Generally, a higher HOMA-B value indicates better beta-cell function, meaning the pancreas is producing insulin effectively.
Time Frame: Visits 5 (week 0), 8 (week 6), and 11 (week 12)
Population: Number of subjects analyzed in the Intent to treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  HOMA-IR Week 6 change from baseline | 0.916 (2.84) | 2.013 (1.943)
  HOMA-IR Week 12 change from baseline | 0.344 (2.32) | -1.833 (3.95)
  HOMA-B Week 6 change from baseline | 12.94 (24.06) | 50.10 (75.81)
  HOMA-B Week 12 change from baseline | -12.41 (38.72) | 47.63 (120.18)

3. Secondary Outcome: Glucose Metabolism HbA1c
Description: Change in HbA1c from Baseline
Time Frame: Visit 5 (week 0), 8 (week 6) and 11 (week 12)
Population: Number of subjects in the Intend to Treat Population who have evaluable results
Measure: Mean (Standard Deviation); unit: percentage of glycated haemoglobin
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 68 | 68
percentage of glycated haemoglobin
  Week 6 change from baseline | 0.02 (0.538) | -0.03 (0.618)
  Week 12 change from baseline | 0.12 (0.659) | 0.03 (0.722)

4. Secondary Outcome: 24 Hours Albumin Excretion
Description: Change in 24 hours Albumin excretion from baseline
Time Frame: Visits 5 (week 0) and 11 (week 12)
Population: Number of subjects analyzed in the intent to treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: mg/24hrs
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 67 | 68
mg/24hrs | 389.82 (1540.30) | -56.15 (1569.23)

5. Secondary Outcome: 24 Hours Urine UACR
Description: Change in 24 hours Urine UACR from baseline
Time Frame: Visits 5 (week 0) and 11 (week 12)
Population: Number of subjects analyzed in the intent to treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 67 | 68
mg/g | 220.15 (592.995) | 169.98 (706.38)

6. Secondary Outcome: eGFR Change by Study Visit
Description: Change in eGFR from baseline by study visit
Time Frame: Visits 5 (week 0), 6 (week 2), 7 (week 4), 8 (week 6), 9 (week 8), 10 (week 10), 11 (week 12), follow up (week 16)
Population: Number of subjects analyzed in the intent to treat Population who have evaluable results
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 68 | 68
mL/min/1.73m^2
  Change in week 2 (Visit 6) eGFR from baseline | -0.5 (6.07) | -0.4 (7.27)
  Change in week 4 (Visit 7) eGFR from baseline | -0.6 (8.25) | -1.5 (6.55)
  Change in week 6 (Visit 8) eGFR from baseline | -0.1 (8.13) | -0.3 (6.80)
  Change in week 8 (Visit 9) eGFR from baseline | -1.1 (8.7) | -1.7 (7.31)
  Change in week 10 (Visit 10) eGFR from baseline | -0.7 (8.21) | -1.9 (7.89)
  Change in week 12 (Visit 11) eGFR from baseline | -1.5 (8.28) | -1.2 (8.08)
  Change in week 16 (Follow up) eGFR from baseline | -1.3 (8.21) | -1.9 (10.45)

7. Other Pre Specified Outcome: Erectile Dysfunction
Description: Changes at week 12 in IEFF questionnaire assessing erectile dysfunction in patients presenting with these diabetic complications at baseline (Baseline <=25 in the erectile function domain)- Score from 1 to 30. Score 1 to 10: severe erectile dysfunction, Score 11-16: moderate erectile dysfunction, Score 17-25: light erectile dysfunction, Score 26-30: normal erectile function
Time Frame: Visits 5 (week 0), and 11 (week 12)
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 46 | 45
score on a scale | 0.8 (5.86) | -0.5 (5.06)

8. Other Pre Specified Outcome: Neuropathic Pain
Description: Changes in Visual Analog Scale (VAS) assessing neuropathic leg pain in patients presenting with these diabetic complications at baseline (subjects with a baseline VAS>=20mm are included). A 100mm VAS scale was used with a range from 0-100mm where a higher score means worse pain. The presence of neuropathic pain is defined a VAS score of at least 20 mm.
Time Frame: Visits 5 (week 0), and 11 (week 12)
Population: Number of subjects analyzed in the Intent to treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GKT137831 | Placebo
Number analyzed (Participants) | 31 | 31
score on a scale | -15.3 (21.79) | -10.5 (22.18)

ADVERSE EVENTS:
Time Frame: Approximately 9-10 months
Description: Adverse events were collected after signing the informed consent form (ICF) and up to completion of the 30-day follow-up period after the last administration of IMP
Arm/Group | GKT137831 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 3/68 | 5/68
Other Adverse Events (participants affected / at risk) | 33/68 | 42/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GKT137831 (N=68) | Placebo (N=68)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Lobular Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GKT137831 (N=68) | Placebo (N=68)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary Tract infection (Infections and infestations) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Edema peripheral (General disorders) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Blood Thyroid Stimulating Hormone increased (Investigations) | 1 (1) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Respiratory, thoracic disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Hypertension (Vascular disorders) | 0 (0) | 2 (3)
Cardiac disorders (Cardiac disorders) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less